CLINICAL TRIAL: NCT03419338
Title: Sinus Lift With Newly Forming Bone and Inorganic Bovine Bone: a Clinical, Histologic and Histomorphometric Evaluation
Brief Title: Sinus Lift With Newly Forming Bone and Inorganic Bovine Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Adriana Campos Passanezi SantAna, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FOBGranSinus
Record Dates: First submitted 2017-10-19; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Maxillary Sinus
Keywords: Maxillary Sinus; Sinus lifting; Bone graft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Surgical alveolus + maxillary sinus lift with inorganic bovine bone + newly forming bone + collagen membrane
  Interventions: Procedure: Sinus lift; Procedure: Surgical alveolus; Procedure: Inorganic bovine bone + newly forming bone; Device: Collagen membrane
- Control group (Active Comparator): Maxillary sinus lift with inorganic bovine bone + collagen membrane
  Interventions: Procedure: Sinus lift; Procedure: Inorganic bovine bone; Device: Collagen membrane

INTERVENTIONS:
Procedure: Sinus lift — Using a lateral access, the Schneider membrane will be elevated using curettes allowing the insertion of graft material.
Procedure: Surgical alveolus — Using a round diamond bur, a surgical alveolus will be created on an toothless ridge region.
  Arms: Test group
Procedure: Inorganic bovine bone + newly forming bone — Maxillary sinus lift will be done with inorganic bovine bone associated with newly forming bone. The newly forming bone will be collected from surgical alveolus previous prepared.
  Arms: Test group
Procedure: Inorganic bovine bone — Maxillary sinus lift will be done with inorganic bovine bone.
  Arms: Control group
Device: Collagen membrane — At the end of the sinus lift, a collagen membrane will be used to obliterate the graft inside the maxillary sinus.

SUMMARY:
The aim of this study is to evaluate the efficacy of newly forming bone graft (NFB) in the gain of bone volume in sinus lift procedures. For that, it will be compared the tomographic bone gain 6 months after surgery between a group that received inorganic bovine bone alone (n=8) and a group that received inorganic bovine bone associated with NFB (n=8).

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of newly forming bone graft (NFB) in the gain of bone volume in sinus lift procedures. It will be recruited for this study individuals 25-60 years of age, both genders, presenting a missing tooth at an upper premolar or molar region with 2-9 mm of remaining bone between alveolar ridge crest and sinus floor and the existence of an edentulous ridge or at least one tooth condemned to extraction. Sinus will be treated by NFB mixed to inorganic bovine bone - IBB (test; n= 8) or IBB (control; n= 8). The volume of bone tissue will be evaluated by computerized tomography obtained at baseline examination and 6 months after surgery. After this period, biopsies of hard tissue will be obtained during implant placement for histologic and histomorphometric analysis.

ELIGIBILITY:
Inclusion Criteria:

• Presenting a distance between alveolar crest and maxillary sinus of 2 to 9 millimeters.

Exclusion Criteria:

* History of periodontal surgery at the area on the last 12 months
* Use of drugs that affect periodontal tissues (eg: anticonvulsants, calcium channel blockers, cyclosporine, bisphosphonates, hormone-based, contraceptives, steroids)
* Pregnant
* Smokers
* Diabetics
* History of head and neck radiotherapy

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Bone height measured in millimeters using the panoramic radiography reconstructions | Six months
  It will be measured the distance between the alveolar ridge and the maxillary sinus in panoramic radiography reconstructions taken before and after sinus lift.

SECONDARY OUTCOMES:
Descriptive histologic analysis of biopsy samples performed by two trained and previously calibrated examiners | Six months
  On the surface and around the particles of the materials with the newformed reactive tissue, it was analyzed the presence and absence of the following tissue and reactive cellular elements: granulation tissue, newly formed blood vessels, fibroblasts, osteoblasts and mineralized bone matrix, foreign body type granuloma, macrophages, inflammatory multinucleated giant cells.
Quantitative histologic analysis of biopsy samples using Leahy et al. (2013) score | Six months
  Quantification of the reactional and reparative phenomena related to cellular and tissue organization on biopsed samples were made using Leahy et al. (2013) score.
Histomorfometric analysis of biopsy samples using percentage of different tissues evaluated at ImageJ | Six months
  The tissue sections were captured with 4x and 10x objective and images were recorded and later analyzed in the ImageJ software. The proportions of vital bone, cortical bone, medullary bone, remnant non-vital particles and connective tissue were quantified separately and expressed as percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana CP Sant'Ana, PhD, Principal Investigator — Bauru School of Dentistry - University of Sao Paulo
Locations (1):
- Bauru School of Dentistry - University of Sao Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided